CLINICAL TRIAL: NCT00658853
Title: Effective High Aerobic Intensity Interval Training to Improve Maximal Oxygen Uptake in COPD Patients
Brief Title: Effective High Aerobic Intensity Endurance Training Regimes in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 149-03
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hyperoxia
Keywords: COPD; training; VO2peak; performance; ventilation; high aerobic intensity treadmill walking; one leg training by cycling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperoxia; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): High aerobic intensity treadmill walking. 4 by 4 minutes interval training on a 5% graded treadmill at a heart rate corresponding to 85-95% of maximal heart rate. 3 times per week for 10 weeks.
  Interventions: Behavioral: 4 times 4 minutes high aerobic intensity one leg cycling
- 2 (Active Comparator): 4 times 4 minutes interval training in hyperoxia - 100% oxygen
  Interventions: Behavioral: 4 times 4 minutes high aerobic intensity one leg cycling
- 3 (Active Comparator): One leg at a time training 4 times 4 minutes interval training using cycling ergometer
  Interventions: Behavioral: 4 times 4 minutes high aerobic intensity one leg cycling

INTERVENTIONS:
Behavioral: 4 times 4 minutes high aerobic intensity one leg cycling — 3 times per week for 10 weeks

SUMMARY:
4 times 4 minutes interval training with and without hyperoxia is more effective than low intensity endurance training.

ELIGIBILITY:
Inclusion Criteria:

* COPD

Exclusion Criteria:

* Heart disease
* Walking or cycling inabilities
* Other diseases

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
VO2peak | 10 weeks
Ventilation | 10 weeks
FEV1 | 10 weeks
Walking performance | 10 weeks

SECONDARY OUTCOMES:
Quality of life | 3 months
SPSS | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Helgerud, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Bjorgen S, Helgerud J, Husby V, Steinshamn S, Richadson RR, Hoff J. Aerobic high intensity one-legged interval cycling improves peak oxygen uptake in chronic obstructive pulmonary disease patients; no additional effect from hyperoxia. Int J Sports Med. 2009 Dec;30(12):872-8. doi: 10.1055/s-0029-1238292. PMID 19821224